CLINICAL TRIAL: NCT05233306
Title: Combined PET and MR Investigations of the Pathophysiology of Gilles de la Tourette Syndrome. Part 2: 7T MRI
Brief Title: Investigations of the Pathophysiology of Gilles de la Tourette Syndrome. Part 2: 7T MRI
Status: Completed | Type: Observational
Sponsor: Max Planck Institute for Human Cognitive and Brain Sciences (Other)
Collaborators: Hannover Medical School (Other); Leipzig University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: PETMR_GTS_2-7T-MRI
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Gilles de la Tourette Syndrome; Tourette Syndrome
Keywords: magnetic resonance imaging; magnetic resonance spectroscopy
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GTS patient group: Cohort of adult GTS patients, males and females, age range 18 to 50 years
  Interventions: Device: MRI scanner (7 Tesla)
- Control group: Cohort of healthy control subjects, males and females, age range 18 to 50 years
  Interventions: Device: MRI scanner (7 Tesla)

INTERVENTIONS:
Device: MRI scanner (7 Tesla) — MRI and MRS examination at 7 Tesla; protocol duration of approx. 75 min

SUMMARY:
Gilles de la Tourette syndrome (GTS; also known as Tourette syndrome) is a congenital neuropsychiatric disorder. Characteristic symptoms are so-called tics-rapid, repetitive movements (motor tics) or vocalizations (vocal tics) that start suddenly without any apparent purpose. Previous research supports the hypothesis of defective regulation (dysregulation) of the dopaminergic system, with particular discussion of dysfunction of tonic/phasic dopamine release or dopaminergic hyperinnervation. Moreover, given the complex interaction of different neurotransmitters, especially in the basal ganglia, it can be assumed that abnormal dopaminergic transmission also affects other transmitter systems, such as glutamate (Glu) or γ-aminobutyrate (GABA). Furthermore, recent results suggest an abnormality in cerebral iron metabolism in GTS. Since iron is accumulated in dopamine vesicles and plays a central role in dopamine synthesis, this observation may also be related to dysfunction of the dopaminergic system. Therefore, in this multimodal study, the investigators aim to combine positron emission tomography (PET), magnetic resonance imaging (MRI), and magnetic resonance spectroscopy (MRS) methods comparing patients with GTS and a control cohort.

In Part 2 of this study, MRI and MRS at 7 Tesla are employed to investigate (i) the concentrations of Glu, glutamine and GABA in the corpus striatum and the cortex cingularis anterior and (ii) the subcortical iron concentration.

DETAILED DESCRIPTION:
State of the Art

Gilles de la Tourette Syndrome (GTS) is characterized by the presence of motor and vocal tics, which have been defined as rapid, habitual, burst-like movements or utterances that typically mimic fragments of normal behavior. Patients often report unpleasant premonitory urge sensations preceding tics that are relieved by their execution. Although the therapeutic spectrum for GTS has recently been expanding, current treatment strategies are often unsatisfactory, thus provoking the need for further elucidation of the underlying pathophysiology.

In current models of GTS pathophysiology, symptoms are thought to arise as a result of the inappropriate activation of specific clusters of striatal neurons, which lead to a burst-like disinhibition of thalamocortical output. The bulk of current literature suggests a dysregulated dopaminergic system. This is supported by clinical evidence of improvements in tics following the administration of dopamine antagonists, synthesis blockers or depletion drugs, and the exacerbation of symptoms following the administration of dopaminergic stimulants. Dopamine drives movement by activating a direct, net excitatory basal ganglia pathway involving the dopamine receptor D1 or an indirect, net inhibitory basal ganglia pathway involving the dopamine receptor D2. Currently, the vast majority of the antipsychotics used for the treatment of tics in GTS aim at the D2 receptor, with aripiprazole, risperidone and pimozide being selective D2 receptor antagonists and haloperidol being mainly a D2 receptor antagonist. However, recent randomized controlled trials further indicate promising results for the selective dopamine receptor D1 antagonist ecopipam.

Methodologically varied work has revealed that patients with GTS exhibit alterations in (i) D2 receptor density or binding, (ii) Dopamine Active Transporter (DAT) density/binding, and (iii) phasic dopamine transmission in striatal and cortical regions. A very small number of post-mortem examinations further suggest potential abnormalities in D1 (and D2 and DAT) receptor densities in cortical regions. While this would be in line with the therapeutic efficiency of selective D1 receptor antagonists, thorough experimental verification is missing. In particular, D1 receptors in GTS patients have not yet been investigated in vivo, suggesting a need for additional research.

Both postsynaptic and presynaptic mechanisms have been postulated to offer explanations of the above observations:

1. Supersensitive postsynaptic dopamine receptors were proposed, in particular to explain findings of reduced levels of homovanillic Acid (HVA) in cerebrospinal fluid (CSF) in GTS despite the premise of a hyperdopaminergic system. The validity of this view has been questioned as HVA levels may be confounded by medication, and previous positron emission tomography (PET) studies on dopamine receptors (although likely involved in the neurobiology of GTS) have produced inconsistent results.
2. Dopamine hyperinnervation, that is, an overabundance of striatal dopamine terminals was suggested to reflect observations of generally increased binding to the DAT and to the vesicular monoamine transporter type 2 (VMAT2).
3. Tonic-phasic dysfunction assumes reduced tonic dopamine levels as well as a hyperresponsive (spike-dependent) phasic dopaminergic system. A low tonic dopamine tone could be caused by an overactive DAT preventing efficient spillage to the extrasynaptic space and/or altered presynaptic dopamine D2 autoreceptor binding.

Apart from such considerations specific to dopamine one can postulate that if a dopaminergic abnormality were present, other neurotransmitter systems would exhibit perturbations as well. In particular, this is suggested by (i) the close synergy exhibited between excitatory, inhibitory and modulatory neurotransmitter systems within the striatum and throughout the brain; and (ii) the interdependent metabolic relationship exhibited between glutamate (Glu), and γ-aminobutyric acid (GABA) via the non-neuroactive metabolic intermediate glutamine (Gln). Moreover, an irregular afferent modulation of dopaminergic nuclei would have profound effects on tonic/phasic dopaminergic release in the striatum and the control of subsequent thalamocortical output. Consistently, separate groups have demonstrated that adult patients with GTS exhibit alterations within the GABAergic system in cortical regions using in vivo proton (1H) magnetic resonance spectroscopy (MRS) and subcortical regions using PET. Employing 1H MRS, the investigators recently found reductions in striatal concentrations of Gln and the sum of Glu plus Gln (Glx) in GTS patients as well as negative correlations between striatal Gln and actual tic severity and between thalamic Glu and premonitory urges. While these findings do not rule out alternative mechanisms, they lend support to the hypothesis of an alteration in the dynamics of the tonic/phasic dopaminergic signaling because chronic perturbations in the subcortical GABA-Glu-Gln cycle flux could lead to spatially focalized alterations in excitatory and inhibitory neurotransmitter ratios.

Another aspect of dopamine neurobiology that has recently gained interest in the context of neuroimaging is the relation to brain iron. Besides supporting myelination and cellular respiration, brain iron is crucial for the synthesis of neurotransmitters, in particular dopamine. It is stored primarily as ferritin and co-localizes with dopamine vesicles having the greatest concentration in the dopamine-rich basal ganglia and midbrain. As the major brain iron compounds have (super)paramagnetic properties, they can be detected via susceptibility-sensitive magnetic resonance (MR) techniques, such as quantitative susceptibility mapping (QSM) or measurements of the effective or the reversible transverse relaxation rates, R2* or R2', respectively. Recent multimodal imaging targeted at (normal) developmental changes of the striatal dopamine system demonstrated that R2'-based estimates of tissue iron content were associated with carbon-11 [11C]dihydrotetrabenazine PET of presynaptic vesicular dopamine. This suggests that susceptibility-sensitive MR imaging (MRI), which does not require an intravenously applied radiotracer, might serve as a proxy for obtaining information on dopamine that could substitute measurements of HVA in CSF without sharing the same confounds. More recently, the investigators already obtained preliminary indications of disturbed iron homeostasis in GTS patients as evidenced by reduced serum ferritin and magnetic susceptibility in the striatum and further subcortical structures.

Objectives and Hypotheses

In continuation of previous investigations, the investigators plan to perform examinations with MRI and MRS in GTS patients in comparison to age- and sex-matched healthy controls within Part 2 of this combined study. This includes (indirect) information on the interplay of different neurotransmitter systems (Glu, and GABA), as well as on the role of brain iron in GTS.

In particular, the investigators plan to use (i) iron-sensitive MRI techniques, such as QSM and R2* mapping; and (ii) 1H MRS with standard single-voxel techniques and spectral-editing methods, for obtaining neurochemical profiles and quantitative information on Glu, Gln, and GABA in the striatum and cortical areas.

Neuropsychological tests:

At the time of the MR and/or PET exams, an established, comprehensive test battery will be performed with all patients for a detailed clinical assessment, including the severity of tics or the presence of comorbidities. These tests may be performed online as a video conference questionnaire and include:

* DSM-IV-symptom list for attention deficit hyperactivity disorder (ADHD), rage attack questionnaire (RAQ), Pittsburgh sleep quality index (PSQI);
* Clinical ratings : Yale global tic severity scale (YGTSS-R), Yale-Brown obsessive-compulsive scale (Y-BOCS), clinical global impression scale (CGI).
* Self-assessment questionnaires: adult tic questionnaire (ATQ), Beck depression inventory (BDI), Beck anxiety inventory (BAI), Conners' adult ADHA rating scales (CAARS), autism spectrum quotient (AQ); premotory urge for tics scale (PUTS), GTS quality of life scale (GTS-QOL).

MR exams within Part 2 (7T MR):

MR scanning at 7 Tesla will be performed to exploit the increased sensitivity available at the higher magnetic field. In particular, this will improve the sensitivity of susceptibility-sensitive MR techniques, which permits to achieve sub-millimeter spatial resolutions for better segmentation of small subcortical structures, such as the subtantia nigra, subthalamic nucleus or red nucleus. Similarly, improved sensitivity and spectral resolution at 7 T will expand the range of accessible metabolites, which allows reliable separation of Glu and Gln as well as improved detectability of GABA. The 7T sub-study comprises the following acquisitions:

* Scout acquisition for automated alignment of imaging or spectroscopy volumes ("auto align").
* Structural MR scan ("MP2RAGE") for image registration, tissue segmentation, morphometry of cortical and subcortical structures, and for measuring the longitudinal relaxation time T1 to obtain information on myelin and brain iron content.
* Susceptibility-sensitive acquisition ("multi-echo FLASH") for measurements of the magnetic susceptibility (QSM) and R2* to obtain information on brain iron and myelin. Note that the MP2RAGE and multi-echo FLASH scans may be combined into a single, simultaneous acquisition of all parameters (susceptibility, T1 and R2*) depending on the results of initial tests in healthy volunteers.
* Single-voxel proton MRS of the basal ganglia and anterior cingulate cortex with both direct and edited acquisitions to obtain concentration estimates of local Glu, Gln, and GABA.

  10ml of venous blood will be collected from all subjects (GTS patients and healthy controls) at the time of the exam for subsequent measurement of blood ferritin levels. These levels will be compared with the results from susceptibility-related measures of brain iron.

ELIGIBILITY:
GTS Group:

Inclusion Criteria:

* GTS according to DSM-IV-TR criteria
* mild or moderate tics
* drug-free for a minimum of 4 weeks prior to the exam

Exclusion Criteria:

* severe tics of the head and/or face
* psychiatric medication within 4 weeks prior to the exam
* consumption of alcohol during 24 hours prior to the exam
* consumption of cannabis during 24 hours prior to the exam
* pregnancy
* general contra-indications for MRI exams

Control Group:

Inclusion Criteria:

* no known neurological or psychiatric disease

Exclusion criteria:

* psychiatric medication within 4 weeks prior to the exam
* consumption of alcohol during 24 hours prior to the exam
* consumption of cannabis during 24 hours prior to the exam
* pregnancy
* general contra-indications for MRI exams

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: GTS group selected from primary care clinic and by advertisement in GTS patient organizations Control group selected from database of the MPI and advertisement
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Subcortical magnetic susceptibility as brain iron proxy | Susceptibility is measured through study completion, an average of 6 months
  Iron stores in subcortical structures are changed in GTS patients
Effective transverse relaxation rate, R2*, as brain iron proxy | R2* is measured through study completion, an average of 6 months
  R2* in subcortical structures is changed in GTS patients
Concentration of glutamate (Glu) and glutamate plus glutamine (Glx) | Glu and Glx are measured through study completion, an average of 6 months
  Glu and Glx levels are changed in GTS patients in striatum and cingulate cortex
Concentration of glutamine (Gln) | Gln is measured through study completion, an average of 6 months
  Gln levels are changed in GTS patients in striatum and cingulate cortex
Concentration of γ-aminobutyrate (GABA) | GABA is measured through study completion, an average of 6 months
  GABA levels are changed in GTS patients in striatum and cingulate cortex

SECONDARY OUTCOMES:
Plasma ferritin level | A plasma sample is analyzed through study completion, an average of 6 months
  Blood ferritin is changed in GTS patients

CONTACTS AND LOCATIONS:
Overall Officials: Harald E Möller, PhD, Principal Investigator — Max Planck Institute for Human Cognitive and Brain Sciences
Locations (1):
- Max Planck Institute for Human Cognitive and Brain Sciences, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kanaan AS, Gerasch S, Garcia-Garcia I, Lampe L, Pampel A, Anwander A, Near J, Moller HE, Muller-Vahl K. Pathological glutamatergic neurotransmission in Gilles de la Tourette syndrome. Brain. 2017 Jan;140(1):218-234. doi: 10.1093/brain/aww285. Epub 2016 Dec 22. PMID 28007998
- [Background] Forde NJ, Kanaan AS, Widomska J, Padmanabhuni SS, Nespoli E, Alexander J, Rodriguez Arranz JI, Fan S, Houssari R, Nawaz MS, Rizzo F, Pagliaroli L, Zilhao NR, Aranyi T, Barta C, Boeckers TM, Boomsma DI, Buisman WR, Buitelaar JK, Cath D, Dietrich A, Driessen N, Drineas P, Dunlap M, Gerasch S, Glennon J, Hengerer B, van den Heuvel OA, Jespersgaard C, Moller HE, Muller-Vahl KR, Openneer TJ, Poelmans G, Pouwels PJ, Scharf JM, Stefansson H, Tumer Z, Veltman DJ, van der Werf YD, Hoekstra PJ, Ludolph A, Paschou P. TS-EUROTRAIN: A European-Wide Investigation and Training Network on the Etiology and Pathophysiology of Gilles de la Tourette Syndrome. Front Neurosci. 2016 Aug 23;10:384. doi: 10.3389/fnins.2016.00384. eCollection 2016. PMID 27601976
- [Background] Albin RL, Mink JW. Recent advances in Tourette syndrome research. Trends Neurosci. 2006 Mar;29(3):175-82. doi: 10.1016/j.tins.2006.01.001. Epub 2006 Jan 23. PMID 16430974
- [Background] Bourne JA. SCH 23390: the first selective dopamine D1-like receptor antagonist. CNS Drug Rev. 2001 Winter;7(4):399-414. doi: 10.1111/j.1527-3458.2001.tb00207.x. PMID 11830757
- [Background] Draper A, Stephenson MC, Jackson GM, Pepes S, Morgan PS, Morris PG, Jackson SR. Increased GABA contributes to enhanced control over motor excitability in Tourette syndrome. Curr Biol. 2014 Oct 6;24(19):2343-7. doi: 10.1016/j.cub.2014.08.038. Epub 2014 Sep 25. PMID 25264251
- [Background] Gilbert DL, Murphy TK, Jankovic J, Budman CL, Black KJ, Kurlan RM, Coffman KA, McCracken JT, Juncos J, Grant JE, Chipkin RE. Ecopipam, a D1 receptor antagonist, for treatment of tourette syndrome in children: A randomized, placebo-controlled crossover study. Mov Disord. 2018 Aug;33(8):1272-1280. doi: 10.1002/mds.27457. Epub 2018 Sep 7. PMID 30192018
- [Background] Kaller S, Rullmann M, Patt M, Becker GA, Luthardt J, Girbardt J, Meyer PM, Werner P, Barthel H, Bresch A, Fritz TH, Hesse S, Sabri O. Test-retest measurements of dopamine D1-type receptors using simultaneous PET/MRI imaging. Eur J Nucl Med Mol Imaging. 2017 Jun;44(6):1025-1032. doi: 10.1007/s00259-017-3645-0. Epub 2017 Feb 14. PMID 28197685
- [Background] Kwak C, Dat Vuong K, Jankovic J. Premonitory sensory phenomenon in Tourette's syndrome. Mov Disord. 2003 Dec;18(12):1530-3. doi: 10.1002/mds.10618. PMID 14673893
- [Background] Larsen B, Olafsson V, Calabro F, Laymon C, Tervo-Clemmens B, Campbell E, Minhas D, Montez D, Price J, Luna B. Maturation of the human striatal dopamine system revealed by PET and quantitative MRI. Nat Commun. 2020 Feb 12;11(1):846. doi: 10.1038/s41467-020-14693-3. PMID 32051403
- [Background] Leckman JF. Tourette's syndrome. Lancet. 2002 Nov 16;360(9345):1577-86. doi: 10.1016/S0140-6736(02)11526-1. PMID 12443611
- [Background] Lerner A, Bagic A, Simmons JM, Mari Z, Bonne O, Xu B, Kazuba D, Herscovitch P, Carson RE, Murphy DL, Drevets WC, Hallett M. Widespread abnormality of the gamma-aminobutyric acid-ergic system in Tourette syndrome. Brain. 2012 Jun;135(Pt 6):1926-36. doi: 10.1093/brain/aws104. Epub 2012 May 10. PMID 22577221
- [Background] Maia TV, Conceicao VA. Dopaminergic Disturbances in Tourette Syndrome: An Integrative Account. Biol Psychiatry. 2018 Sep 1;84(5):332-344. doi: 10.1016/j.biopsych.2018.02.1172. Epub 2018 Mar 9. PMID 29656800
- [Background] Mink JW. Basal ganglia dysfunction in Tourette's syndrome: a new hypothesis. Pediatr Neurol. 2001 Sep;25(3):190-8. doi: 10.1016/s0887-8994(01)00262-4. PMID 11587872
- [Background] Moller HE, Bossoni L, Connor JR, Crichton RR, Does MD, Ward RJ, Zecca L, Zucca FA, Ronen I. Iron, Myelin, and the Brain: Neuroimaging Meets Neurobiology. Trends Neurosci. 2019 Jun;42(6):384-401. doi: 10.1016/j.tins.2019.03.009. Epub 2019 Apr 29. PMID 31047721
- [Background] Okubo Y, Suhara T, Suzuki K, Kobayashi K, Inoue O, Terasaki O, Someya Y, Sassa T, Sudo Y, Matsushima E, Iyo M, Tateno Y, Toru M. Decreased prefrontal dopamine D1 receptors in schizophrenia revealed by PET. Nature. 1997 Feb 13;385(6617):634-6. doi: 10.1038/385634a0. PMID 9024661
- [Background] Singer HS. Treatment of tics and tourette syndrome. Curr Treat Options Neurol. 2010 Nov;12(6):539-61. doi: 10.1007/s11940-010-0095-4. PMID 20848326
- [Background] Singer HS, Morris C, Grados M. Glutamatergic modulatory therapy for Tourette syndrome. Med Hypotheses. 2010 May;74(5):862-7. doi: 10.1016/j.mehy.2009.11.028. Epub 2009 Dec 21. PMID 20022434
- [Background] Tinaz S, Belluscio BA, Malone P, van der Veen JW, Hallett M, Horovitz SG. Role of the sensorimotor cortex in Tourette syndrome using multimodal imaging. Hum Brain Mapp. 2014 Dec;35(12):5834-46. doi: 10.1002/hbm.22588. Epub 2014 Jul 15. PMID 25044024
- [Background] Yoon DY, Gause CD, Leckman JF, Singer HS. Frontal dopaminergic abnormality in Tourette syndrome: a postmortem analysis. J Neurol Sci. 2007 Apr 15;255(1-2):50-6. doi: 10.1016/j.jns.2007.01.069. Epub 2007 Mar 6. PMID 17337006